CLINICAL TRIAL: NCT03871023
Title: The Use of Prophylactic Negative Wound Therapy in Emergency and Elective Laparotomy Wounds
Brief Title: Prophylactic Negative Wound Therapy in Laparotomy Wounds.
Acronym: PROPEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Noel Edward Donlon, Specialist Registrar General Surgery, St. James's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SJH0519
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Wound Infection; Wounds; Dehisence; Cosmesis; Home Care; Length of Hospital Stay
MeSH Terms: conditions — Wound Infection; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 3 separate treatment arms
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Simple dressing (Active Comparator): Standard, waterproof dressing applied to wound
  Interventions: Device: Smith & Nephew PICO Negative wound pressure versus standard dresing; Device: PREVENA Negative pressure wound versus standard dressing
- PICO Dressing (Active Comparator): Negative Wound pressure applied second cohort
  Interventions: Device: PREVENA Negative pressure wound versus standard dressing
- PREVENA Dressing (Active Comparator): Negative wound presure applied to third cohort
  Interventions: Device: Smith & Nephew PICO Negative wound pressure versus standard dresing

INTERVENTIONS:
Device: Smith & Nephew PICO Negative wound pressure versus standard dresing — To investigate if negative wound pressure improves wound outcome
  Arms: PREVENA Dressing; Simple dressing
Device: PREVENA Negative pressure wound versus standard dressing — To investigate if negative wound pressure improves wound outcome
  Arms: PICO Dressing; Simple dressing

SUMMARY:
Post-operative wound issues in abdominal surgery have a significant impact on patient outcomes. The impact of different types of wound therapy are not clear in the literature.

The hypothesis of this study is that NPWT has the potential to reduce Surgical Site Infections, however no study has compared the most commonly used products against standard dressings.

DETAILED DESCRIPTION:
In the era of enhanced recovery, improving modifiable peri-operative and post-operative factors is essential to better patient outcomes. Surgical site complications in the form of wound infections are a major burden to the healthcare system. Negative pressure wound therapy (NPWT) as delivered by a surgical incision management system (SIMS) is a novel approach to improve wound healing when applied to closed incisions.

However, data is limited in its application to laparotomy incisions in the acute and elective care surgery setting. Surgical site infections can complicate a patient's post-operative course significantly, often necessitating a longer length of stay, antibiotic therapy, intervention for wound collections and impair patient mobility and overall recovery.

In addition to this, laparotomy wound complications can possibly delay adjuvant therapy and also increases healthcare costs both as an inpatient and in the community. Despite significant measures to reduce such complications in the form of wound care bundles, changing of gloves prior to wound closure etc, surgical site complications continue to represent a huge healthcare burden.

Aim;

1. To determine if prophylactic negative pressure wound therapy confers a lower rate of Superficial Site Infection or reduces wound complications in Emergency or Elective Laparotomy wounds thereby improving post-operative patient recovery and reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 years of age undergoing a laparotomy are eligible for entry into this study. Benign and malignant conditions are eligible for inclusion.

Exclusion Criteria:

* Pregnant patients and those undergoing re-look laparotomies are to be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-11-06 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
superficial site infection via southampton scoring system (higher score - worse outcome) | 5 days
  seroma/haematoma/abscess formation
Wound Dehisence | 5 days
  disruption of wound continuity

SECONDARY OUTCOMES:
Wound healing/Cosmesis | week 6 post op
  scar healing (via observer scar assesment scale - higher score wore outcome)
Length of hospital stay | 30 days
  wound complications causing prolonged hospital stay
home care therapy | 30days
  lenth of home care dressings

CONTACTS AND LOCATIONS:
Overall Officials: Noel E Donlon, Principal Investigator — St. James's Hospital, Ireland
Locations (1):
- St. James' Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Deleted post analysis

REFERENCES:
- [Derived] Donlon NE, Boland PA, Kelly ME, Schmidt K, Cooke F, Neary PM, Barry KM, Reynolds JV. Prophylactic negative wound therapy in laparotomy wounds (PROPEL trial): randomized controlled trial. Int J Colorectal Dis. 2019 Nov;34(11):2003-2010. doi: 10.1007/s00384-019-03398-9. Epub 2019 Sep 16. PMID 31529194